CLINICAL TRIAL: NCT00809536
Title: A Phase 1, Open-Label, Randomized, Cross-Over Study To Estimate The Pharmacokinetics Of PD 0332334 And Metformin When Administered Concurrently In Healthy Subjects
Brief Title: Investigation Of How PD 0332334 And Metformin Are Eliminated From The Body When They Are Administered At The Same Time
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Please Detailed Description for termination reason.
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: A5361031
Record Dates: First submitted 2008-12-15; First posted 2008-12-17 (Estimated); Last update posted 2010-02-17 (Estimated); Status verified 2010-02

CONDITIONS: Generalized Anxiety Disorder
Keywords: metformin, PD 0332334, organic cation transporter, OCT2, pharmacokinetics
MeSH Terms: conditions — Generalized Anxiety Disorder | interventions — Metformin; imagabalin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1 (Other): This is an open-label, randomized, two period cross-over which will be conducted in 12 healthy adults
  Interventions: Drug: Metformin
- Cohort 2 (Other): This is an open-label, randomized, two period cross-over which will be conducted in 12 healthy adults
  Interventions: Drug: PD 0332334

INTERVENTIONS:
Drug: Metformin — 225 mg q12, oral PD 0332334 immediate release formulation on Days 1 through 5; Single, oral, 500 mg dose of metformin immediate release
  Other Names: imagabalin
  Arms: Cohort 1
Drug: Metformin — Single, oral, 500 mg of metformin immediate release
  Arms: Cohort 1
Drug: PD 0332334 — 500 mg q12, oral metformin immediate release administered on Days 1 through Day 6 Single, oral, 300 mg dose of PD 0332334 immediate release formulation administered on Day 3
  Arms: Cohort 2
Drug: PD 0332334 — Single, oral, 300 mg dose of PD 0332334 immediate release formulation
  Arms: Cohort 2

SUMMARY:
1. To estimate the effects of multiple doses of PD 0332334 on the elimination of a single dose of metformin from the body
2. To estimate the effects of multiple doses of metformin on the elimination of a single dose of PD 0332334 from the body
3. To evaluate the safety and tolerability when PD 0332334 and metformin are administered at the same time.

DETAILED DESCRIPTION:
Detailed Description:

Additional Study Purpose Details: To assess the pharmacokinetics of metformin and PD 0332334 with concurrent administration.

On February 18th 2009, a decision to terminate further development for PD 0332334 was communicated to investigators in this study. The decision to terminate this study was not based on any safety concerns.

ELIGIBILITY:
Inclusion Criteria:

* Nonsmokers
* Male or female adults

Exclusion Criteria:

* Current or history of significant medical illness
* Smokers
* Illicit drug use

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2009-01; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Metformin and PD 0332334 area under the curve (AUC) from time 0 to infinity (AUCinf) | Days 1 through 7
Metformin and PD 0332334 AUC from 0 to last quantifiable concentration (AUClast) | Days 1 through 7
Metformin and PD 0332334 half-life (t1/2) | Days 1 through 7
Metformin and PD 0332334 maximum plasma concentration | Days 1 through 7

SECONDARY OUTCOMES:
Clinical safety laboratories | Days 1 through 7
Incidence, duration and severity of adverse events when study medications administered alone and concurrently | Days 1 through 7
Discontinuation due to adverse events when study medications administered alone and concurrently | Days 1 through 7
12-lead ECGs | Days 1 through 7
Vital signs | Days 1 through 7

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Singapore, Singapore

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5361031&StudyName=Investigation%20Of%20How%20PD%200332334%20And%20Metformin%20Are%20Eliminated%20From%20The%20Body%20When%20They%20Are%20Administered%20At%20The%20Same%20Time